CLINICAL TRIAL: NCT04332575
Title: Clinical Extend Study to Evaluate Safety and Effectiveness of TnR Nasal Mesh for Correction of Nasal Septum on Patients Who Need Correction of Nasal Septum That Accompanies With Rhinanchone Symptom
Brief Title: Clinical Extend Study to Evaluate Safety and Effectiveness of TnR Nasal Mesh for Correction of Nasal Septum on Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: T&R Biofab Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRBF-002
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Septal Deformity; Nasal Obstruction
Keywords: Nasal obstruction; Septal deformity; Septoplasty; TnR Nasal Mesh; polycaprolactone
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observation study is to evaluate long term safety and efficacy at 2~3 years after surgery on patients who have completed nasal septal deformity surgery using TnR Nasal Mesh.

DETAILED DESCRIPTION:
Nasal obstruction is a nasal disease commonly seen in the area of otolaryngology, and major symptoms include nasal congestion, rhinitis, and etc.

Nasal septoplasty is a surgery performed to improve above symptoms of nasal obstruction and so far, many surgical technique have been studied. All surgical techniques aimed to improve breathing through the nasal cavity by supporting the end of nose using surgical materials such as autologous bone or nonabsorbable material.

In the case of autologous bone transplantation, safety is ensured, but there is a limitation since it causes deficiency of the donor site, and the nasal septum may be altered by a modification of the implanted tissue.

In the case of nonabsorbable materials, there is a high risk of side effects such as hyposmia, septal perforation, and occurrence of boil.

TnR Nasal Mesh, as a surgical material for nasal septoplasty has a sufficient flexural strength to support the nasal septum and to overcome the force of returning to a deviated state prior to surgery.

Animal tests have shown that TnR Nasal mesh well supports the nasal septum after surgery and the surrounding tissue is well fused between the pores without inflammatory responses. Based on above results, a clinical trial was planned to evaluate long term safety and efficacy of TnR Nasal Mesh as a material for nasal septoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have completed nasal septal deformity surgery using TnR Nasal Mesh.
2. Females of childbearing potential must have a negative urine pregnancy test, and must not plan to become pregnant during the course of the study.
3. A person who voluntarily signed a consent form after hearing and understanding the description of this clinical study.

Exclusion Criteria:

1. Pregnancy or lactation

   * Before screening
2. History of surgery in nasal or paranasal sinuses before screening
3. History of radiation treatment at Head and neck
4. History of having participated in other clinical trial of a drug/ a medical device within three months

   * Screening point
5. Patients with untreated nasal bone fraction or trauma of nasal
6. Patients with surgical site infection caused by nasal bone fraction or trauma
7. Patients with inflammation in a nasal cavity
8. Patients with asthma
9. Patients with untreated a perforation of septum, a sinusitis, a nasal cavity polyposis, a nasal cavity sarcoidosis, nasal valve collapse or wegener's granulomatosis
10. Patients with sarcoma or carcinoma in a nasal cavity
11. Patients with untreated palate-facial disfigurements or cleft palate
12. Patients with sepsis
13. Patients with systemic inflammatory disease
14. Patients who are unsuitable for clinical sturdy determined by the researcher.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 19 and 74, who have completed nasal septal deformity surgery using TnR Nasal Mesh.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Total NOSE score change after surgery compared to before surgery | 1 day
  The descriptive statistics(population, mean, standard deviation, median, minimum, maximun value) are presented for total NOSE score change after surgery compared to before surgery.
  All measurement will be completed at the time of each patient's initial visit, 1 day
  Total NOSE score of before surgery is based on the results of previous clinical study.
  The NOSE(Nasal Obstruction Symptom Evaluation) score is a 5-step scale (0(asymptomatic)-4(very severe) points) of the severity of each symptom over the past month for the 5 symptoms related to nasal obstruction (nasal hyperemia / snagging / difficulty in breathing / sleeping disorder / difficulty breathing during exercise). Then, it is evaluated by interviewing patient. The total score of 20 points is converted to 100 points and recorded.

SECONDARY OUTCOMES:
NOSE score change | 1 day
  NOSE score change for each item after surgery compared to before.
  All measurement will be completed at the time of each patient's initial visit, 1 day
  The NOSE(Nasal Obstruction Symptom Evaluation) score is a 5-step scale (0(asymptomatic)-4(very severe) points) of the severity of each symptom over the past month for the 5 symptoms related to nasal obstruction (nasal hyperemia / snagging / difficulty in breathing / sleeping disorder / difficulty breathing during exercise). Then, it is evaluated by interviewing the patient. The total score of 20 points is converted to 100 points and recorded.
Acoustic rhinometry results(volume) | 1 day
  Changes after surgery compared to before surgery on bilateral nasal cavity volume in acoustic rhinometry result.
  All measurement will be completed at the time of each patient's initial visit, 1 day
Acoustic rhinometry results(cross sectional area) | 1 day
  Changes after surgery compared to before surgery on bilateral nasal cavity cross sectional area in acoustic rhinometry result.
  All measurement will be completed at the time of each patient's initial visit, 1 day
CT images(cross sectional area) | 1 day
  Changes after surgery compared to before surgery on bilateral nasal cavity cross sectional area in CT images.
  All measurement will be completed at the time of each patient's initial visit, 1 day
CT images(ratio of convex to concave side) | 1 day
  Changes after surgery compared to before surgery on nasal cavity ratio of convex to concave side of cross-sectional area in CT images.
  All measurement will be completed at the time of each patient's initial visit, 1 day
CT images(nasal septum angle) | 1 day
  Changes after surgery compared to before surgery on nasal septum angle in CT images.
  All measurement will be completed at the time of each patient's initial visit, 1 day
Ratio of improvement of regarding symptoms after surgery | 1 day
  Symptom improvement is defined as the total NOSE score reduced by more than 40 points compared to before surgery or the total NOSE score less than 20 points after surgery.
  All measurement will be completed at the time of each patient's initial visit, 1 day
  The NOSE(Nasal Obstruction Symptom Evaluation) score is a 5-step scale (0(asymptomatic)-4(very severe) points) of the severity of each symptom over the past month for the 5 symptoms related to nasal obstruction (nasal hyperemia / snagging / difficulty in breathing / sleeping disorder / difficulty breathing during exercise). Then, it is evaluated by interviewing the patient. The total score of 20 points is converted to 100 points and recorded.
Level of satisfaction of patients using VAS | 1 day
  The patient satisfaction is evaluated using VAS(Visual Analogue Scale).
  All measurement will be completed at the time of each patient's initial visit, 1 day
  VAS(Visual Analogue Scles)Scoring and Interpretation Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-won Kim, professor, Study Director — The Catholic University of Korea

REFERENCES:
- [Background] Surowitz J, Lee MK, Most SP. Anterior Septal Reconstruction for Treatment of Severe Caudal Septal Deviation: Clinical Severity and Outcomes. Otolaryngol Head Neck Surg. 2015 Jul;153(1):27-33. doi: 10.1177/0194599815582176. Epub 2015 Apr 16. PMID 25883105
- [Background] Kim JH, Kim DY, Jang YJ. Outcomes after endonasal septoplasty using caudal septal batten grafting. Am J Rhinol Allergy. 2011 Jul-Aug;25(4):e166-70. doi: 10.2500/ajra.2011.25.3648. PMID 21819753
- [Background] Rimmer J, Ferguson LM, Saleh HA. Versatile applications of the polydioxanone plate in rhinoplasty and septal surgery. Arch Facial Plast Surg. 2012 Sep-Oct;14(5):323-30. doi: 10.1001/archfacial.2012.147. PMID 22986938
- [Background] Boenisch M, Nolst Trenite GJ. Reconstruction of the nasal septum using polydioxanone plate. Arch Facial Plast Surg. 2010 Jan-Feb;12(1):4-10. doi: 10.1001/archfacial.2009.103. PMID 20083734
- [Background] Kahveci OK, Miman MC, Yucel A, Yucedag F, Okur E, Altuntas A. The efficiency of Nose Obstruction Symptom Evaluation (NOSE) scale on patients with nasal septal deviation. Auris Nasus Larynx. 2012 Jun;39(3):275-9. doi: 10.1016/j.anl.2011.08.006. Epub 2011 Aug 31. PMID 21885221
- [Background] Stewart MG, Smith TL, Weaver EM, Witsell DL, Yueh B, Hannley MT, Johnson JT. Outcomes after nasal septoplasty: results from the Nasal Obstruction Septoplasty Effectiveness (NOSE) study. Otolaryngol Head Neck Surg. 2004 Mar;130(3):283-90. doi: 10.1016/j.otohns.2003.12.004. PMID 15054368
- [Background] Kim JN, Choi HG, Kim SH, Park HJ, Shin DH, Jo DI, Kim CK, Uhm KI. The efficacy of bioabsorbable mesh as an internal splint in primary septoplasty. Arch Plast Surg. 2012 Sep;39(5):561-4. doi: 10.5999/aps.2012.39.5.561. Epub 2012 Sep 12. PMID 23094256
- [Background] Garcia LB, Oliveira PW, Vidigal Tde A, Suguri Vde M, Santos Rde P, Gregorio LC. Caudal septoplasty: efficacy of a surgical technique-preliminary report. Braz J Otorhinolaryngol. 2011 Mar-Apr;77(2):178-84. doi: 10.1590/s1808-86942011000200007. PMID 21537619
- [Background] Erickson B, Hurowitz R, Jeffery C, Ansari K, El Hakim H, Wright ED, Seikaly H, Greig SR, Cote DW. Acoustic rhinometry and video endoscopic scoring to evaluate postoperative outcomes in endonasal spreader graft surgery with septoplasty and turbinoplasty for nasal valve collapse. J Otolaryngol Head Neck Surg. 2016 Jan 12;45:2. doi: 10.1186/s40463-016-0115-9. PMID 26754620
- See also: Description SIDS Initial Assessment Report — http://webnet.oecd.org/hpv/UI/handler.axd?id=2ccdc186-93a9-47cd-b91d-26789738233d